CLINICAL TRIAL: NCT03338049
Title: Multicenter, Prospective Trial of ElectromagnetIc Bronchoscopic and Electromagnetic Transthoracic Navigational Approaches for the Biopsy of Peripheral Pulmonary Nodules
Brief Title: All in One Study: A Prospective Trial of Electromagnetic Navigation for Biopsy of Pulmonary Nodules
Acronym: AIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Veran Medical Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: VMT AIO 2017
Record Dates: First submitted 2017-10-25; First posted 2017-11-09 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Veran System (Other): Staged biopsy sampling methodology. If lymph node staging is negative, EMN-bronchoscopy will be performed. If EMN-bronchoscopy is negative, EMN-TTNA will be performed
  Interventions: Device: Veran System

INTERVENTIONS:
Device: Veran System — Electromagnetic navigation bronchoscopy and electromagnetic navigation transthoracic needle aspiration
  Other Names: Veran SPiN Thoracic Navigation System SPiNPerc Kit

SUMMARY:
This is a multi-center, non-randomized, single-arm, prospective trial to evaluate a staged sampling methodology designed to maximize the diagnostic yield of lung biopsy in a single procedure setting.

DETAILED DESCRIPTION:
The objectives of this study are to evaluate diagnostic yield following biopsy of peripheral pulmonary nodules as identified on chest computed tomography (CT) utilizing (1) Electromagnetic navigation (EMN) bronchoscopy, and/or (2) EMN-transthoracic needle aspiration (TTNA). Overall diagnostic yield will be evaluated to assess the combination of these approaches.

ELIGIBILITY:
Inclusion Criteria:

* The patient is ≥21 years old,
* The patient has a lung nodule identified on chest CT and is a candidate for elective EMN bronchoscopic evaluation as determined by the treating pulmonologist,
* The size of the target nodule, as measured at its greatest diameter, is between 1-3cm,
* Staging at the time of enrollment indicates NO/N1 (does not involve lymph nodes or includes involvement in nodes within ipsilateral hilum),
* The patient has an intermediate risk of malignancy (5-65% per the Mayo Model) and is in need of diagnosis for alternative treatment, OR The patient has a high probability of cancer (>65%) and will be referred for surgical evaluation or stereotactic body radiation therapy (SBRT). Note: If the patient refuses surgery or if the surgeon requests a definitive diagnosis prior to surgery the patient will have the option to be included in this study,
* The patient has a lack of bleeding disorders, and
* The patient is willing and able to provide informed consent.

Exclusion Criteria:

* The patient is pregnant as confirmed by urine or serum pregnancy testing,
* The patients has a body mass index (BMI) >40,
* There is a predetermined plan to pursue stereotactic body radiation therapy (SBRT) in the event of a nondiagnostic study procedure in patients with a nodule within SPiNPerc range (i.e. The patient would not go on for a CT guided TTNA), OR There is a predetermined plan to pursue stereotactic body radiation therapy (SBRT) in the event of a nondiagnostic study procedure in patients where the target nodule is within a region considered to be not accessible to a percutaneous approach as determined by the radiology core lab and thus would prevent a confirmatory tissue diagnosis before SBRT.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2019-10-29 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic Yield | Up to one year post index procedure
  Diagnostic yield associated with either EMN-bronchoscopy or EMN-TTNA

SECONDARY OUTCOMES:
Serious Adverse Events | 30 days post index procedure
  All device and/or procedure related serious adverse events
Adverse Events | 30 days post index procedure
  Rate of all device and procedure related events
Rate of procedure cancellation | On procedure day
  Impact of same day CT scan on rate of procedure cancellations due decrease in nodule size
Procedural Factors | Intra-procedure
  Number of instrument passes, type of instrument, site of biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Lonny Yarmus, DO, Principal Investigator — Johns Hopkins University
Locations (9):
- United States (9):
  - Banner University Medical Center - Phoenix, Phoenix, Arizona
  - Grady Memorial Hospital, Atlanta, Georgia
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Washington University Medical Center, St Louis, Missouri
  - University of North Carolina Medical Center, Chapel Hill, North Carolina
  - Duke University Hospital, Durham, North Carolina
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina Medical Center, Charleston, South Carolina
  - Swedish Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thiboutot J, Pastis NJ, Akulian J, Silvestri GA, Chen A, Wahidi MM, Gilbert CR, Lin CT, Los J, Flenaugh E, Semaan R, Burks AC, Sathyanarayan P, Wu S, Feller-Kopman D, Cheng GZ, Alalawi R, Rahman NM, Maldonado F, Lee HJ, Yarmus L. A Multicenter, Single-Arm, Prospective Trial Assessing the Diagnostic Yield of Electromagnetic Bronchoscopic and Transthoracic Navigation for Peripheral Pulmonary Nodules. Am J Respir Crit Care Med. 2023 Oct 15;208(8):837-845. doi: 10.1164/rccm.202301-0099OC. PMID 37582154
- [Derived] Mallow C, Lee H, Oberg C, Thiboutot J, Akulian J, Burks AC, Luna B, Benzaquen S, Batra H, Cardenas-Garcia J, Toth J, Heidecker J, Belanger A, McClune J, Osman U, Lakshminarayanan V, Pastis N, Silvestri G, Chen A, Yarmus L. Safety and diagnostic performance of pulmonologists performing electromagnetic guided percutaneous lung biopsy (SPiNperc). Respirology. 2019 May;24(5):453-458. doi: 10.1111/resp.13471. Epub 2019 Jan 24. PMID 30675961
- [Derived] Thiboutot J, Lee HJ, Silvestri GA, Chen A, Wahidi MM, Gilbert CR, Pastis NJ, Los J, Barriere AM, Mallow C, Salwen B, Dinga MJ, Flenaugh EL, Akulian JA, Semaan R, Yarmus LB. Study Design and Rationale: A Multicenter, Prospective Trial of Electromagnetic Bronchoscopic and Electromagnetic Transthoracic Navigational Approaches for the Biopsy of Peripheral Pulmonary Nodules (ALL IN ONE Trial). Contemp Clin Trials. 2018 Aug;71:88-95. doi: 10.1016/j.cct.2018.06.007. Epub 2018 Jun 7. PMID 29885373